CLINICAL TRIAL: NCT06463847
Title: Single Center, Open-label, Dose-increasing Phase I Clinical Trial of UC-MSCs for the Treatment of Knee Osteoarthritis
Brief Title: Phase I Clinical Trial of UC-MSCs in the Treatment of Knee Osteoarthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Hamilton Biotechnology Co., Ltd (Unknown); Guangzhou Hamilton Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UHCT240051
Record Dates: First submitted 2024-04-22; First posted 2024-06-18 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; UC-MSCs; Cell Therapy; Safety; DLT; Efficiency
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1UC-MSCs Treatment Group (Experimental): Participants will receive conventional treatment plus 1 time of UC-MSCs (5×10^6 UC-MSCs/2.5mL, single injection into the knee cavity).
  Interventions: Drug: UC-MSCs
- 2UC-MSCs Treatment Group (Experimental): Participants will receive conventional treatment plus 1 time of UC-MSCs (1×10^7 UC-MSCs/2.5mL, single injection into the knee cavity).
  Interventions: Drug: UC-MSCs
- 3UC-MSCs Treatment Group (Experimental): Participants will receive conventional treatment plus 1 time of UC-MSCs (2×10^7 UC-MSCs/2.5mL, single injection into the knee cavity).
  Interventions: Drug: UC-MSCs

INTERVENTIONS:
Drug: UC-MSCs — In this study, three dose groups are preset, which are low-dose group: 5×10^6 cells/2.5mL; medium-dose group: 1×10^7 cells/2.5mL; high-dose group: 2×10^7cells/2.5mL, 9 to 18 subjects will be recruited, and will be sequential from the low-dose group to the high-dose group according to the "3+3" dose escalation principle. At least 3 subjects are enrolled in each group for the safety and tolerability test of single administration. After the last subject in each dose group completes the DLT observation period, the sponsor and the researcher jointly confirm the safety tolerance of the subjects in the previous dose group, and only after the safe tolerance is determined can the subjects enter the next dose group, so as to evaluate the safety and tolerance of human umbilical cord mesenchymal stem cell injection in the treatment of knee osteoarthritis. Recommend appropriate cell therapy dose (RP2D) for Phase II clinical trials.

SUMMARY:
In recent years, the incidence rate and disability rate of osteoarthritis have continued to grow, and it has become a common chronic disease of elderly patients, second only to the "three highs", and poses a continuous threat to China's medical and health system and public health system. Knee osteoarthritis is the main type of osteoarthritis, ranking 11th in global disability diseases and 38th in disability adjusted life year loss, causing significant economic burden to patients, families, and society. At present, most of the treatment methods for KOA have limited efficacy, only relieving pain symptoms and cannot prevent cartilage damage and other tissue damage in the joints. Due to the limitations of adverse events, there is still no optimal treatment plan for KOA. Most studies believe that autologous mesenchymal stem cell transplantation is a new treatment method with good efficacy and good repair effect for mild to moderate cartilage defects. Given that there is currently no optimal treatment plan for KOA, human umbilical cord mesenchymal stem cell injection has potential development value and is of great significance for the treatment of KOA patients.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic inflammatory disease of the bone and joints, characterized by degenerative destruction of articular cartilage, subchondral bone sclerosis and osteophyte formation, and peripheral soft tissue inflammation and proliferation. Knee Osteoarthritis (KOA), which is negative and highly active, is the most common. Currently, there are approximately 1 billion KOA patients worldwide, with approximately 150 million patients in China, and the incidence rate increases with age. The clinical manifestation of KOA is repeated and prolonged bone and joint pain, which seriously affects the patient's quality of life, ultimately leading to joint structural damage and loss of function, causing a significant burden on individuals, families, and society. At present, there is a lack of effective treatment methods for KOA both domestically and internationally, and there is an urgent need to research new treatment strategies to meet clinical needs. Numerous studies have shown that local inflammation of the joint cavity and apoptosis of articular chondrocytes are the main pathological mechanisms of knee osteoarthritis. Therefore, the key to treating KOA is to inhibit the local inflammatory response of bone joints, promote chondrocyte regeneration, repair damaged joint surfaces, and restore their normal structure and function.

Mesenchymal Stem Cells (MSCs) are the most widely studied pluripotent stem cells. It exists in various tissues, has multidirectional differentiation potential, homing effect and powerful paracrine function, can regulate tissue microenvironment, promote damaged tissue repair through cell replacement, promote in-situ cell regeneration, anti-inflammatory and immune regulation and other mechanisms. Therefore, mesenchymal stem cell therapy has become the focus of KOA new therapy research. A large number of studies have shown that MSCs can be induced to differentiate into stable mature chondrocytes that can express proteoglycan and type II collagen. Fluorescently labeled MSCs could still be detected 10 weeks after injection into the joint cavity of osteoarthritis model animals, suggesting that MSCs homed in the injured articular cartilage tissue and participated in the regeneration and repair of the injured tissue. The effectiveness of MSCs therapy for KOA has been demonstrated in osteoarthritis models in different animals including rats, rabbits, sheep, pigs, and monkeys. MSCs from different sources can effectively inhibit the inflammatory response and chondrocyte injury in model animals, and stimulate the regeneration and repair of injured chondrocytes.

In this study, three dose groups are preset, which are low-dose group: 5×10^6 cells/2.5mL; medium-dose group: 1×10^7 cells/2.5mL; high-dose group: 2×10^7cells/2.5mL, 9 to 18 subjects will be recruited, and will be sequential from the low-dose group to the high-dose group according to the "3+3" dose escalation principle. At least 3 subjects are enrolled in each group for the safety and tolerability test of single administration. After the last subject in each dose group completes the DLT observation period, the sponsor and the researcher jointly confirm the safety tolerance of the subjects in the previous dose group, and only after the safe tolerance is determined can the subjects enter the next dose group, so as to evaluate the safety and tolerance of human umbilical cord mesenchymal stem cell injection in the treatment of knee osteoarthritis. Recommend appropriate cell therapy dose (RP2D) for Phase II clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Prior to conducting any assessment, written informed consent must be obtained;
* Able to communicate well with researchers during screening, understand and comply with experimental requirements;
* Age range from 50 to 70 years old (including threshold), regardless of gender;
* Male weight ≥ 50 kg, female weight ≥ 45 kg, body mass index (BMI) within the range of 18-26 kg/m2 (including critical values);
* According to the diagnostic criteria for knee osteoarthritis in the "Guidelines for the Diagnosis and Treatment of Osteoarthritis (2018 Edition)", subjects diagnosed with knee osteoarthritis (see Annex 1 for details); The course of knee osteoarthritis is more than 4 weeks;
* The target knee joint X-ray Kellgren Lawrence radiological grading (K-L IV grade) is II-III grade. Patients diagnosed with knee osteoarthritis on both sides should have non target knee joint symptoms, signs, and grading that do not exceed the target knee joint;
* MRI examination shows partial or full layer damage to the cartilage of the knee joint;
* A VAS score of ≥ 5 and ≤ 7 for knee joint pain at least 48 hours after discontinuing the use of all painkillers during screening;
* Patients who use analgesic therapy (taking paracetamol/acetaminophen) to control local pain in the target knee joint agree to discontinue the use of similar analgesics 2 weeks prior to administration, and only allow NSAID as a rescue drug; Patients who use glucosamine, chondroitin, opioid drugs, or diacetate, glucosamine, etc. must agree to discontinue such drugs from 2 weeks prior to administration.

Exclusion Criteria:

* Individuals with a history of knee joint infection, surgery, and radiation therapy within 6 months prior to administration;
* Combined instability of the knee joint (anterior and posterior cruciate ligaments, medial and lateral collateral ligaments), rupture, relaxation, or external deformity of the knee joint;
* According to researchers, diseases that may interfere with knee joint function assessment, such as symptomatic lower back pain, lumbar disc herniation, and hip joint pain in the target knee joint;
* According to the judgment of researchers, local diseases that may confuse knee joint function assessment include but are not limited to septic arthritis, reactive arthritis, clinically recurrent pseudogout, chondrocalcinosis, or joint fractures;
* Within 3 months prior to administration, any medication injection treatment (including intra-articular injection of growth factors, hormones, or sodium hyaluronate) or lavage surgery has been received in the knee joint (target side) cavity;
* Merge intra-articular or periarticular tumors (such as knee synovial chondroma, pigmented nodular synovitis, etc.);
* Various serious systemic diseases such as neurological disorders, respiratory disorders, heart diseases (NYHA grade III and above), and liver dysfunction (ALT>3) × ULN or AST>3 × ULN, renal dysfunction (Cr>2) × ULN or BUN>2 × ULN, coagulation dysfunction (INR>1.5), or severe hematological disorders (such as grade 3 or above anemia, hemoglobin (Hb)<8 g/dL, grade 2 or above thrombocytopenia, PLT<75) × 10 ^ 9/L);
* Diagnosed as systemic inflammatory arthritis or connective tissue disease, including but not limited to rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, gout, Paget's disease, systemic lupus erythematosus, or other systemic diseases that may confuse KOA assessment (such as fibromyalgia);
* Subjects who receive long-term (>14 days) oral corticosteroids>5 mg/day within 3 months prior to administration, or who require long-term glucocorticoid treatment during the trial period;
* Previously received stem cell therapy;
* Uncontrolled hypertension is defined as systolic blood pressure (SBP)>160 mmHg or diastolic blood pressure (DBP)>100 mmHg during screening;
* Having a history of tumors, mental illness, severe autoimmune diseases, hematological diseases, and long-term use of immunosuppressants;
* Have a history of alcohol and prohibited drug abuse;
* Has a history of hypersensitivity to protein drugs;
* There are contraindications to MRI examination or unwillingness to undergo MRI examination;
* Hepatitis B, hepatitis C, AIDS, syphilis serological test positive pathogens;
* Pregnant or lactating women, or male or female patients who tested positive for blood pregnancy during screening or have planned childbirth within 3 months after medication;
* Patients who have received live vaccines or attenuated live vaccines within one month before administration;
* Patients who have participated in clinical trials of other drugs or devices within 3 months prior to administration;
* Patients with poor compliance, poor communication skills, inability to adhere to follow-up, and inability to complete the entire trial;
* The researchers believe that it is not suitable for participants to enter this experiment.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | From Baseline (0 W) to 4 weeks after treatment
  Incidence and severity of adverse events after administration (CTCAE 5.0)

SECONDARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities Arthritis Index，with the minimum value 0, and the maximum value 240, and higher scores mean a worse outcome) | From Baseline (0 W) to 24 hours, 4 weeks, 12 weeks, 24 weeks, 48 weeks after treatment
  Changes in WOMAC score from baseline
VAS (Visual Analogue Scale,with the minimum value 0, and the maximum value 10, and higher scores mean a worse outcome) | From Baseline (0 W) to 24 hours, 4 weeks, 12 weeks, 24 weeks, 48 weeks after treatment
  Changes in VAS score from baseline
Changes in knee joint range of motion from baseline | From Baseline (0 W) to 4 weeks, 12 weeks, 24 weeks, 48 weeks after treatment]
  Changes in knee joint range of motion from baseline
Changes in X-Kellgren-Lawrence grading and minimum joint space width (mJSW) from baseline | From Baseline (0 W) to 24 weeks, 48 weeks after treatment
  Changes in X-Kellgren-Lawrence grading and minimum joint space width (mJSW) from baseline
Changes of MRI-Roberts cartilage repair score, cartilage thickness and synovial inflammation score (reference MOAKS) compared with baseline | From Baseline (0 W) to 24 weeks, 48 weeks after treatment
  MRI-Roberts score includes cartilage repair score, cartilage thickness and synovial inflammation score，with different grades according to the situation，and the higher grades mean a worse situation (reference MOAKS（Magnetic Resonance imaging Osteoarthritis Knee Score），but not all indicators of MOAKS are included)

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China